CLINICAL TRIAL: NCT05982522
Title: A Multicenter, Open-Label, Randomized, Phase Ib/II Clinical Trial to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of IN10018 Combined With Taxane and Anti-PD-1/L1 Monoclonal Antibody in Previously-treated Solid Tumors
Brief Title: IN10018 Combination Therapy in Previously-treated Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-017
Record Dates: First submitted 2023-07-13; First posted 2023-08-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): IN10018 + nab-paclitaxel + Tislelizumab in previously-treated NSCLC
  Interventions: Drug: IN10018; Drug: Nab-paclitaxel; Drug: Tislelizumab
- Control Group (Active Comparator): Nab-paclitaxel + Tislelizumab in previously-treated NSCLC
  Interventions: Drug: Nab-paclitaxel; Drug: Tislelizumab

INTERVENTIONS:
Drug: IN10018 — orally taken once daily
  Other Names: BI 853520
  Arms: Experimental Group
Drug: Nab-paclitaxel — 125 mg/m2 D1, 8 Q3W, Intravenously
Drug: Tislelizumab — 200mg Q3W, Intravenously

SUMMARY:
This is a phase Ib/II, randomized, open-label, multicenter clinical trial to evaluate the antitumor activities, safety, tolerability and pharmacokinetics (PK) of IN10018 in combination with taxane and anti-PD-1/L1 monoclonal antibody in patients with locally advanced or metastatic solid tumors who have failed in or been intolerant to at least one line of standard therapy. This study will be firstly carried out in previously-treated non-small cell lung cancer (NSCLC) population,

DETAILED DESCRIPTION:
This study consists of 2 parts: 1) Phase Ib-Dose Confirmation part: To assess the safety and recommended phase II dose (RP2D) of IN10018 in combination with taxane (nab-paclitaxel is proposed) and anti-PD-1/L1 monoclonal antibody (Tislelizumab is proposed) in previously-treated solid tumors. 2) Phase II-Dose Expansion part: To assess the antitumor efficacy and safety of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors. This study will be firstly carried out in previously-treated NSCLC population, and after getting enough efficacy and safety data of IN10018+nab-paclitaxel+Tislelizumab in NSCLC population and also taken into consideration of disease background of other specific solid tumors, sponsor will decide if to expand the treatment regimen into other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years old at the time of signing informed consent.
2. Be able to understand and be willing to sign informed consent.
3. Histologically or cytologically confirmed NSCLC, which is not suitable for locallly radical therapy.

   Note: Subjects should have received prior platinum-based doublet chemotherapy and anti-PD-1/L1-based systemic therapy and failed in treatment.
4. Subjects who have failed in 1- to 2 prior lines of standard systemic therapy.
5. Has at least one measurable tumor lesion per RECIST 1.1.
6. Has an ECOG performance status of 0 or 1.
7. Estimated life expectancy is more than 3 months.
8. Has adequate organ function.
9. AEs due to prior antitumor therapy must be recovered to ≤ Grade 1 (CTCAE v5.0) or a steady state as assessed by investigators
10. Subjects (male and female) with childbearing potential must agree to use contraception during the treatment phase and through 3 months after the last dose of study treatment.

Exclusion Criteria:

1. Previously documented EGFR, ALK and ROS1 mutation.
2. Have received chemotherapy, biological therapy, endocrine therapy, immunotherapy and other antitumor drugs within 4 weeks prior to the first dose of study treatment.
3. Have received other antitumor investigational drugs or treatments within 4 weeks prior to the first dose of study treatment.
4. Have received radiotherapy within 14 days prior to the first dose of study treatment.
5. Have had allogeneic haematopoietic stem cell transplantation or organ transplantation.
6. History of autoimmune disease within the past 2 years.
7. Have an immunodeficiency disorder or have received systemic steroid therapy (prednisone or equivalent corticosteroid > 10 mg/day) or other immunosuppressants within 7 days prior to the first dose of study treatment.
8. Currently have interstitial pneumonitis.
9. Have had FAK inhibitors treatment.
10. Have received prior nab-paclitaxel treatment and the first documented disease progression/recurrence is within 6 months since the last dose of nab-paclitaxel treatment.
11. Malignancies other than the study disease within 3 years prior to the first dose of study treatment.
12. Active central nervous system (CNS) metastases and/or carcinogenic meningitis.
13. Has a history of severe cardiovascular or cerebrovascular diseases within 6 months prior to the first dose.
14. Pleural, pericardial or abdominal effusion that are clinically symptomatic and require puncture or drainage.
15. Any active infection requiring systemic therapy within 14 days prior to the first dose of study treatment.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study. Note: Subjects who have experienced Grade ≥ 3 immuno-related AEs (irAEs) during prior immunotherapy will not be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-13 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of IN10018 in combination with nab-paclitaxel and Tislelizumab | 3 years
  Evaluate the number of patients with dose-limited toxicities (DLTs); Determine the RP2D of IN10018 in combination with nab-paclitaxel and Tislelizumab.
Objective response rate (ORR) of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors per blinded independent central review (BICR) based on RECIST 1.1 | 3 years
  Defined as the proportion of subjects with complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors per BICR and investigators based on RECIST 1.1 | 3 years
  Defined as the time from randomization to first documentation of disease progression or to death due to any cause, whichever comes first.
Duration of objective response (DOR) of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors per BICR and investigators based on RECIST 1.1 | 3 years
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
Disease Control Rate (DCR) of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors per BICR and investigators based on RECIST 1.1. | 3 years
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
Objective response rate (ORR) of IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors per investigators based on RECIST 1.1. | 3 years
  Defined as the proportion of subjects with complete response (CR) or partial response (PR).
Overall survival (OS) in IN10018+nab-paclitaxel+Tislelizumab as compared to nab-paclitaxel+Tislelizumab in previously-treated solid tumors. | 3 years
  Defined as the time from randomization to the date of death due to any cause.
Number of patients with adverse event | 3 years
  The number of participants who experienced AEs is presented.
PK: AUC of IN10018 following single dose administration and at steady state | 3 years
  Area under the concentration-time curve (AUC)
PK: Cmax of IN10018 following single dose administration and at steady state | 3 years
  Maximum concentration (Cmax)
PK:Ctrough of IN10018 following single dose administration and at steady state | 3 years
  Trough concentration (Ctrough)
PK:Tmax of IN10018 following single dose administration and at steady state | 3 years
  Time to Cmax (Tmax)
PK:t1/2 of IN10018 following single dose administration and at steady state | 3 years
  Elimination half-life (t1/2).
PK:CL/F of IN10018 following single dose administration and at steady state | 3 years
  apparent clearance (CL/F)
PK:Vd/F of IN10018 following single dose administration and at steady state | 3 years
  Apparent volume of distribution (Vd/F)

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, Principal Investigator — Jiangsu Province Cancer Hosipital

IPD SHARING:
Plan to Share IPD: No